CLINICAL TRIAL: NCT06586697
Title: Sequential Thoracic Radiotherapy for Extensive-stage Small-cell Lung Cancer Treated with Chemo-immunotherapy Followed by PD-1/PD-L1 Inhibitor Maintenance Therapy：a Phase II, Single Arm, Prospective Trial
Brief Title: First-line Treatment for ES-SCLC with Chemotherapy Combined with PD-1/PD-L1 Inhibitor Sequential Thoracic Radiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC-II-01
Record Dates: First submitted 2024-05-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thoracic Radiotherapy (Experimental): Thoracic Radiotherapy (45Gy /1.5Gy/bid/3w)
  Interventions: Radiation: Thoracic Radiotherapy

INTERVENTIONS:
Radiation: Thoracic Radiotherapy — Thoracic Radiotherapy (45Gy /1.5Gy/bid/3w)

SUMMARY:
This is an open-label, single arm Phase II study designed to observe and evaluate the efficacy and safety of sequential thoracic radiotherapy in the first-line treatment of extensive small cell lung cancer with chemotherapy combined with approved PD-1/PD-L1 inhibitors.

DETAILED DESCRIPTION:
This study a single arm prospective phase II study. All the enrolled patients will be patients with ES-SCLC who did not have PD after 4-6 cycle of platinum-based chemotherapy in combination with an PD-1/PD-L1 inhibitors. Then, those enrolled patients would be treated with thoracic radiotherapy concurrently with PD-1/PD-L1 maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between18 years and 75 years.
2. Histologic or cytologic confirmation of extensive-stage small cell lung cancer.
3. Initially treated patients with extensive SCLC showed no disease progression after 4-6 cycles of chemotherapy combined with PD-1/PD-L1 inhibitors.
4. Presence of at least one measurable lesion (according to RECIST v1.1).
5. ECOG performance status of 0 or 1.
6. Life expectancy of at least 3 months.
7. Adequate bone marrow, liver and kidney function.
8. Adequate pulmonary function with FEV1 >1 L or >30 % of predicted value and DLCO >30 % of predicted value

Exclusion Criteria:

1. Previous T cell co-stimulation or immune checkpoint therapy.
2. Previous received chemoradiotherapy for limited-stage SCLC.
3. Central nervous system metastasis with clinical symptoms.
4. Multiple liver metastases (patients with isolated liver metastases, metastatic lesions < 3cm could be included).
5. Patients with spinal cord compression.
6. Idiopathic pulmonary fibrosis, institutional pneumonia, drug-induced pneumonia or idiopathic pneumonia, or evidence of active pneumonia during screening (patients with active pulmonary tuberculosis couldn't be enrolled).
7. Have received any other investigational drug treatment or participated in another interventional clinical study within 4 weeks prior to signing the informed consent.
8. In the 5 years prior to the study, subjects had prior or concurrent malignancies requiring active treatment.
9. Subjects with any severe and/or uncontrolled disease (hypertension, heart disease, infection, cirrhosis, active hepatitis, AIDS, third space effusion).
10. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
11. Severe allergic reactions to any of the monoclonal antibodies are known to occur.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate at 6-month | 12 months after last patient entry
  PFS is defined as the period from the start of receiving the first line chemotherapy plus PD-1/PD-L1 inhibitor to disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- HenanCH, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No